CLINICAL TRIAL: NCT06775366
Title: Effects of General Anesthesia with Remimazolam and Propofol on Rhythmic State and Cognitive Function
Brief Title: The Effect of General Anesthesia with Remimazolam and Propofol on Rhythmic State and Cognitive Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RPPOCD
Record Dates: First submitted 2025-01-01; First posted 2025-01-15 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Functioning; Propofol; Remimazolam; Circadian Rhythm
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- remimazolam for general anesthesia (Experimental): Remimazolam 6mg/kg/h was pumped intravenously for 2.5 min, Sufentanil 0.5 μg/kg and rocuronium 0.6mg/kg were injected intravenously, and endotracheal intubation was performed 3 minutes later. Remimazolam was then pumped at 1 mg/kg/h, the BIS was kept in the range of 40-60 through general anesthesia, and the remimazolam infusion rate was adjusted (0.5-3 mg/kg/h).If the BIS cannot be maintained at ≤ 60 or there are signs of potential inadequate anesthesia (such as cough, sweating, and patient movement), and the maximum infusion dose of remimazolam has been given, supplemental sedation with the remedial drug sevoflurane or propofol is used and the case is dismissed.
  Interventions: Drug: Remimazolam
- propofol for general anesthesia (Active Comparator): Propofol (2-3mg/kg), Sufentanil (0.5μg /kg), rocuronium (0.6mg/kg) were injected intravenously, and endotracheal intubation was performed for 3 minutes. Subsequently, propofol was pumped at 4-10mg/kg/h to maintain the BIS in the range of 40-60.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam 6mg/kg/h was pumped intravenously for 2.5 min, Sufentanil 0.5 μg/kg and rocuronium 0.6mg/kg were injected intravenously, and endotracheal intubation was performed 3 minutes later. Remimazolam was then pumped at 1 mg/kg/h, the BIS was kept in the range of 40-60 through general anesthesia, and the remimazolam infusion rate was adjusted (0.5-3 mg/kg/h).If the BIS cannot be maintained at ≤ 60 or there are signs of potential inadequate anesthesia (such as cough, sweating, and patient movement), and the maximum infusion dose of remimazolam has been given, supplemental sedation with the remedial drug sevoflurane or propofol is used and the case is dismissed.
  Arms: remimazolam for general anesthesia
Drug: propofol — Propofol (2-3mg/kg), Sufentanil (0.5μg /kg), rocuronium (0.6mg/kg) were injected intravenously, and endotracheal intubation was performed for 3 minutes. Subsequently, propofol was pumped at 4-10mg/kg/h to maintain the BIS in the range of 40-60.
  Arms: propofol for general anesthesia

SUMMARY:
This study want to observe the effects of remimazolam and propofol for general anesthesia on postoperative rhythm and cognitive function. The observation group was given remimazolam for general anesthesia, and the control group was given propofol for general anesthesia. Both drugs are commonly used as intravenous anesthetics for general anesthesia and have been shown to be safe for use in general anesthesia. The investigators hope can understand the effects of remimazolam and propofol for general anesthesia on rhythm status and cognitive function through this study, further reduce the occurrence of postoperative cognitive function impairment, and enable subjects to better recover.

DETAILED DESCRIPTION:
Benzodiazepines are one of the most important and commonly used intravenous sedatives in the perioperative period. However, benzodiazepines are often associated with a variety of side effects, including respiratory depression, cardiovascular depression, excessive sedation, delayed recovery, disturbance of consciousness, dizziness and nausea, postoperative delirium, and postoperative cognitive impairment. Remimazolam is a new type of benzodiazepine anesthetic drug. It can be rapidly hydrolyzed into inactive carboxylic acid metabolites by widely existing carboxylesterases in the human body. Therefore, it has the characteristics of fast onset, fast metabolism, little impact on liver and kidney function, and little inhibition of respiratory circulation. However, as a benzodiazepine, remimazolam has little effect on postoperative cognitive function.

Biorhythms are currently a hot topic in medical research. Many organisms, including mammals, have the suprachiasmatic nucleus (SCN), a circadian clock pacemaker located in the hypothalamus, which drives the rhythms of activity and rest, fasting and eating, body temperature and hormones to synchronize to 24 hours. Many anesthetic drugs, such as propofol, dexmedetomidine, and volatile anesthetic drugs such as sevoflurane and desflurane, interfere with the expression of circadian rhythm genes in mammals. For example, the expression of rhythm genes per1 and per2 in supratasmatic nucleus of rats injected with a single dose of propofol is down-regulated, and irregular resting activity rhythm is observed in patients undergoing colonoscopy under anesthesia with propofol. The circadian period of patients undergoing general anesthesia is obviously advanced, and the disturbance of circadian rhythm is an important feature of postoperative sleep disorders. However, sleep disorders can aggravate postoperative delirium and postoperative cognitive dysfunction, and related rhythm genes such as Dbp participate in the plasticity of the hippocampus, so the interference of anesthesia drugs on the biological rhythm of the body may be an important cause of postoperative cognitive dysfunction. Since propofol is commonly used in clinical intravenous anesthesia, this study intends to compare the effects of remimazolam and propofol on patients' activity rest rhythm and their effects on learning and memory functions.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years old, ASAI-III class, BMI18.5-25kg/m2 Inpatients undergoing laparoscopic cholecystectomy The estimated time of operation is 1.5~2.5 hours Preoperative brief mental status examination (MMSE) score ≥24 Voluntary participation and signed informed consent

Exclusion Criteria:

Pregnant or lactating women Patients who are allergic to remimazolam or contraindicated Patients who are dependent on or tolerant to opioids or have long-term alcoholism Serious cardiovascular system, respiratory system, liver and kidney diseases History of obstructive sleep apnea mental disorders or neurological diseases Patients who participated in clinical trials of other drugs within the last 3 months The attending physician or researcher considers that there are other circumstances that are not suitable for participation in this study Refuse to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | 30 minutes after extubation and 24 hours after surgery
  The digital symbol task was measured 30 minutes after extubation and 24 hours after surgery to assess the patient's attention and executive ability. The test requires subjects to quickly transcribe numbers into symbols within their line of sight. The score is the number of correct numeric symbols recorded by the subject within 20 seconds.
Cognitive function | 30 minutes after extubation and 24 hours after surgery
  The finger tap test was measured 30 minutes after extubation and 24 hours after surgery to assess the fine motor ability. The average stroke number of a normal person within a 10-second time limit is about 40, and the speed of the right hand is about 1.1 times that of the left hand. The test includes a keystroke and a device that records the number of keystrokes. We performed this test using a tablet: a square area was placed in the middle of the screen to allow the subject to click as quickly as possible, while the tablet automatically recorded the completion time.The subjects were asked to complete 10 seconds of tapping with each hand separately and take short breaks between each test.Record the number of strokes each hand completes in 10 seconds.
Cognitive function | 30 minutes after extubation and 24 hours after surgery
  The digital span test was measured 30 minutes after extubation and 24 hours after surgery to assess the short-term memory. The digital span test assays memory ability and attention span by having subjects recall the correct number immediately after seeing a randomly appearing string of numbers and input it into an electronic device, and increase the length of the string one digit at a time after remembering it correctly. Record the length of the numeric string that the subject can eventually recall.
Cognitive function | 30 minutes after extubation and 24 hours after surgery
  The stroop color word test was measured 30 minutes after extubation and 24 hours after surgery to assess the distraction and conditioned reflex suppression. Mixing words with different colors and meanings and the same meaning in the center of the screen (for example, on the word "green" written in red) requires subjects to quickly select the meaning of the word and suppress automatic reflexes to recognize the color. Record the subject completion time.
Cognitive function | 30 minutes after extubation and 24 hours after surgery
  The schulte square test was measured 30 minutes after extubation and 24 hours after surgery to assess the patient attention level ability. The investigators used a tablet to do this test: there are 16 grids in the center of the screen. The grid is arbitrarily filled with Arabic numerals 1-16, with a total of 16 digits. During the test, participants were asked to manually click on number locations in order of 1-16, and only after clicking the correct location could they proceed to the next number click. The software automatically records the time spent. Subjects were asked to complete two trials each time, with a short break between each trial, and to record the shortest time to complete the trial between the two tests.

SECONDARY OUTCOMES:
Patient activity/rest condition | 30 minutes after extubation and 24 hours after surgery
  From 24 hours before surgery to 24 hours after surgery, the patient will wear a Huawei sports bracelet to record the patient's activity and rest condition
The quality of recovery score | 24 hours after surgery to complete the QoR-15 score assessment
  The quality of postoperative recovery was assessed by quality of recovery score-15(QoR-15). The quality of postoperative recovery score includes 15 questions, with a maximum of 10 points for each question, a maximum of 150 points, and a minimum of 0 points. The higher the score, the better the patient's recovery quality.
ramsay sedation score | 30min after extubation to complete the ramsay sedation score assessment
  The degree of sedation was assessed by ramsay sedation score.1 score: restlessness;2 points: sober, quiet and cooperative;3 points: lethargy, quick response to instructions;4 points: light sleep state, can quickly wake up;5 points: sleep, slow response to calls;6 points: Deep sleep, unresponsive to calls.
Anesthesia adverse events | during surgery
  such as hypotension, hypertension, bradycardia or other anesthesia adverse events
drug-related adverse reactions | during surgery
  Adverse reactions, such as respiratory depression, itching, coughing, irritability, drowsiness, dizziness, delirium, or other adverse reactions
Use of vasoactive drugs | during surgery
  The use of vasoactive drugs during the operation was recorded
fluid volume | during surgery
  Record the Infusion volume during the surgery
Record the time of extubation | From the end of the surgery to leaving the postoperative recovery room
  Record the time of extubation
Numerical rating scale 24 hours after surgery | from 24 hours after surgery to complete the NRS pain assessment
  The degree of postoperative pain was assessed by the numerical rating scale(NRS). A minimum score of 0 means no pain. A maximum score of 10 represents the highest level of pain.
Postoperative nausea numerical rating scale | from 24 hours after surgery to complete the postoperative nausea NRS score
  The degree of postoperative nausea was assessed by the nausea numerical rating scale. A minimum score of 0 means no nausea. The highest score of 10, represents the most intense nausea.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 2024.11---2026.11